CLINICAL TRIAL: NCT04827446
Title: A Randomized Trial Of The SYNC APP
Brief Title: Lighting Intervention for Cancer-related Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Arcascope, Inc (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UMCC 2020.157; HUM00191617 (Other: UM IRB); R44CA236557 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Prostate Cancer; Hematologic Malignancy; Survivorship; Fatigue
Keywords: Fatigue; light therapy; mobile app
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Hematologic Neoplasms; Fatigue

STUDY DESIGN:
Intervention Model Description: Blocked randomization will be used to limit bias and achieve an equal distribution of participants to the intervention and control arms of the study (69 control, 69 intervention; with 23 from each cancer population in each arm). This approach will recruit participants in small blocks to ensure that half of the participants within each block will be allocated to the treatment and the other half to the control.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Light intervention delivered through SYNC app + blue-light blocking glasses.
  Interventions: Other: Wearable Sensor; Other: Blue-blocking glasses; Other: Full SYNC app
- Control Arm (Active Comparator): Placebo light intervention delivered through SYNC app + clear glasses.
  Interventions: Other: Wearable Sensor; Other: Clear glasses; Other: "Dummy" SYNC app

INTERVENTIONS:
Other: Wearable Sensor — Patient is given a wearable device to wear for 12 weeks.
  Other Names: Apple Watch or Fitbit Charge 3
Other: Blue-blocking glasses — Patient is given blue-blocking glasses to wear at instructed times.
  Arms: Intervention Arm
Other: Clear glasses — Patient is given glasses that block no visible light.
  Arms: Control Arm
Other: Full SYNC app — Patient downloads the SYNC app and is given light interventions designed to have a targeted, personalized effect on the circadian clock.
  Arms: Intervention Arm
Other: "Dummy" SYNC app — Patient downloads the SYNC app and is given light interventions designed to have minimal impact on the circadian clock.
  Arms: Control Arm

SUMMARY:
Fatigue is a major problem for cancer patients, and one that can persist long after treatment ends. Recent work has demonstrated that light therapy may mitigate or reduce fatigue levels in both cancer patients and cancer survivors. This protocol seeks to assess how lighting interventions distributed through a mobile app affect fatigue, sleep, and quality of life across three populations of cancer patients: breast cancer and prostate cancer, and patients who have undergone autologous hematopoietic stem cell transplant (HSCT). Participants will be randomized 1:1 to either the interventional SYNC app or to a control app.

ELIGIBILITY:
Inclusion Criteria

* Must own an iPhone 6s or later (with iOS 14 or later or willing to update to iOS 14+) and be willing to complete surveys on it, per the protocol.
* Sleep aid usage will be allowed as long as the patient has been on a stable dose for at least 4 weeks prior to enrollment and agrees to continue the same dose during the study.
* A response of at least 4 on a 10 point scale (with 0 = not fatigued at all and 10 = extremely fatigued) to the question "How fatigued did you feel in the past week?"
* Breast cancer population: Diagnosed with stage 1-3 breast cancer in the last 10 years, without metastatic disease. Chemotherapy or radiation therapy, if indicated, must have been completed at least 3 months prior to enrollment. Concomitant anti-HER2 therapy and/or anti-endocrine therapy is permitted.
* Prostate cancer population: Undergoing androgen deprivation therapy (ADT) for at least three months and are anticipated to remain on ADT for the duration of the trial. Concomitant additional anti-androgen therapy (e.g., enzalutamide) is permitted.
* Autologous HSCT population: Participants must be from the University of Michigan Blood and Marrow Transplant Program.

Exclusion Criteria

* The patient cannot be undergoing chemotherapy at the time of enrollment, but post transplant maintenance therapy that begins after enrollment is allowed.
* The patient must have no evidence of disease progression or recurrence. Specifically for the prostate cancer population, the patient must have no evidence of disease progression on their current ADT regimen at the time of enrollment.
* The patient must not be a night shift worker, where night shift is defined as working a significant number of hours (i.e. more than half) between the hours of 11PM and 6AM on a regular basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Choi, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayer C, Walch O, Dempsey W, Hannay K, Clingan C, Bowen Z, Rozwadowski M, Reichert ZR, Henry NL, Alumkal JJ, Tewari M, Forger DB, Choi SW. A circadian and app-based personalized lighting intervention for the reduction of cancer-related fatigue. Cell Rep Med. 2025 Mar 18;6(3):102001. doi: 10.1016/j.xcrm.2025.102001. Epub 2025 Mar 7. PMID 40056908
- See also: Related Info — http://www.arcascope.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 70 | 69
Completed | 65 | 66
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Customized [Mean (Full Range); unit: years] — Population: Separated by arm and cancer population
  years
    Breast: number analyzed (Participants) | 23 | 23 | 46
    Breast | 52.09 [33 to 72] | 57 [41 to 74] | 54.55 [33 to 74]
    Prostate: number analyzed (Participants) | 21 | 21 | 42
    Prostate | 70.24 [50 to 87] | 67.24 [51 to 76] | 68.74 [50 to 87]
    HSCT: number analyzed (Participants) | 21 | 22 | 43
    HSCT | 54.95 [19 to 74] | 53.91 [25 to 73] | 54.43 [19 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 30 | 31 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 60 | 64 | 124
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 60 | 59 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 65 | 66 | 131

OUTCOME MEASURES:

1. Primary Outcome: Change in Fatigue Assessed With Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) Fatigue 4a
Description: The primary outcome was PROMIS® Fatigue 4a Short Form (SF) at the end of trial, compared between arms. As we did not have a PROMIS® 4-item Fatigue weekly measurement for week 0, we were unable to calculate a change from baseline through this measure alone. We assessed this outcome by looking at differences in fatigue between the intervention and control group at the final week (week 11), and the treatment effect on fatigue at week 11 while controlling (through generalized estimating equations) for baseline fatigue with the 1-item Fatigue question ("In the past 7 days, how would you rate your fatigue on average?") taken from the pre-trial PROMIS® Global Health survey. The 1-item question about fatigue on the pre and post-trial Global Health surveys was scored on a scale from 0 (least fatigued) to 4 (most fatigued).
Time Frame: 11 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 66
score on a scale
  Week 1 fatigue T-scores | 2.18 (0.68) | 2.03 (0.53)
  Week 11 fatigue T-scores | 1.70 (0.74) | 1.58 (0.61)

2. Secondary Outcome: Change in Level of Sleep Disturbance Using PROMIS SF Sleep Disturbance 8a
Description: 8-item PROMIS sleep disturbance questionnaire completed on the first day and last day of the patient's time on study. Each item is on a scale of 1 - 5, best (1) to worst (5). Mean scores are to be compared between the pre-trial and post-trial assessments. A higher score indicates more severe sleep disturbance. The T-Score metric is used to convert the raw score to a standard score, the T-score represents a standardized measure of sleep disturbance, with a mean of 50 and a standard deviation of 10.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 66
T Score
  Pre-trial | 55.84 (6.81) | 53.71 (6.29)
  Post- Trial | 51.85 (6.31) | 52.06 (6.03)

3. Secondary Outcome: Change in Level of Anxiety Using PROMIS SF Anxiety 7a
Description: 7-item PROMIS anxiety questionnaire completed on the first day and last day of the patient's time on study. Each item is on a scale of 1 - 5, best (1) to worst (5). Mean scores are to be compared between the pre-trial and post-trial assessments. A higher score indicates greater anxiety levels. The T-Score metric is used to convert the raw score to a standard score and the range is around 36-74 with a mean score around 50.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 66
T Score
  Pre-trial | 53.16 (9.06) | 51.71 (7.73)
  Post-trial | 50.54 (8.98) | 50.93 (7.17)

4. Secondary Outcome: Change in Level of Depression Using PROMIS SF Depression 8a
Description: 8-item PROMIS depression questionnaire completed on the first day and last day of the patient's time on study. Each item is on a scale of 1 - 5, best (1) to worst (5). Mean scores are to be compared between the pre-trial and post-trial assessments. A higher score indicates greater severity of depression. The T-Score metric is used to convert the raw score to a standard score and a typical range is around 40-60. T-scores are standardized, with a mean of 50 and a standard deviation of 10
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 66
T Score
  Pre-trial | 50.94 (7.55) | 49.90 (6.76)
  Post-trial | 49.25 (8.25) | 48.03 (6.75)

5. Secondary Outcome: Change in Level of Physical Function Using PROMIS SF Physical Function 8b
Description: 8-item PROMIS physical function questionnaire completed on the first day and last day of the patient's time on study. Each item is on a scale of 1 - 5, best (1) to worst (5). Mean scores are to be compared between the pre-trial and post-trial assessments. A higher score indicates better physical function. The T-Score metric is used to convert the raw score to a standard score. The T-score has a mean of 50 and a standard deviation of 10
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 66
T Score
  Pre-Trial | 43.25 (8.20) | 45.07 (8.03)
  Post- Trial | 44.66 (8.31) | 46.40 (7.71)

6. Secondary Outcome: Change in Overall Health Metrics Using PROMIS Global-10
Description: PROMIS Global-10 is a 10-question survey used as an overall evaluation of one's physical and mental health. Mean scores are to be compared between the pre-trial and post-trial assessments for both physical and mental health. A higher score indicates better overall health. The T-Score metric is used to convert the raw score to a standard score and a typical range is 0-100. The T-score has a mean of 50 and a standard deviation of 10
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 66
T Score
  Pre-trial Physical Health | 41.67 (5.66) | 42.82 (4.45)
  Post-trial Physical Health | 42.96 (5.76) | 44.16 (4.81)
  Pre-trial Mental Health | 46.24 (7.45) | 47.61 (6.37)
  Post-trial Mental Health | 47.31 (8.06) | 47.38 (6.51)

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were not collected as part of this trial. All Cause Mortality was assessed over a period of 2 years
Description: Adverse Events and Serious Adverse Events were not collected as part of this trial. All Cause Mortality was assessed over a period of 2 years
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 2/65 | 4/66
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT04827446/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04827446/ICF_000.pdf